CLINICAL TRIAL: NCT03939039
Title: Genetical Characterization of Patients Presenting With Dyslipidemia
Brief Title: From Known to New Genes in Dyslipidemia
Acronym: GENELIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: GENELIP
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Deoxyribonucleic Acid (DNA) of patients will sequenced using Sanger and Illumina Next-Generation Sequencing (NGS) methodology combined with PapilLyon, the pipeline developed by the Hospices Civils de Lyon (HCL) bioinformatics team, which allows more than 350 genes potentially involved in plasma lipoprotein metabolism to be explored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dyslipidemia: Genotype/phenotype correlation in patients with dyslipidemia

SUMMARY:
The mechanism of the majority of the dyslipidemia is multifactorial at the molecular level and remains elusive in more than 50% of the patients in many clinical conditions. Next generation sequencing, a booming strategy, improves the molecular diagnosis efficiency in both monogenic and polygenic dyslipidemia.

In order to decipher the mechanisms involved in the occurrence of dyslipidemia, in addition to the exploration of known candidate genes and Single Nucleotide Polymorphisms (SNP) involved in polygenic modulation, new genes involved in the regulation of lipoprotein metabolism or associated with lipids concentrations need to be sequenced in large groups of dyslipidemic patients.

The goal of this project is to gain new insight into genotype/phenotype correlation.

ELIGIBILITY:
Inclusion Criteria:

* patients with a family documented history of primary hypercholesterolemia, hypertriglyceridemia, hypobetalipoproteinemia, combined hypolipidemia and combined hyperlipidemia according to the European Atherosclerosis Society and/or published data.
* patients with major secondary dyslipidemia.

Exclusion Criteria:

* inability to provide written informed consent
* lack of legal representative

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Male or female patients with dyslipidemia
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2000-01-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Genetical exploration in dyslipidemic patients | 25 years
  Deoxyribonucleic Acid (DNA) sequencing will allow the study of rare gene variants and their frequency in known and new genes in patients with dyslipidemia.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Moulin, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Laboratoire de Biologie Médicale Multi Sites, Centre de Biologie et de Pathologie Est, Département de biochimie et biologie moléculaire Grand Est, Bron, France

REFERENCES:
- [Derived] Vanhoye X, Bardel C, Rimbert A, Moulin P, Rollat-Farnier PA, Muntaner M, Marmontel O, Dumont S, Charriere S, Cornelis F, Ducluzeau PH, Fonteille A, Nobecourt E, Peretti N, Schillo F, Wargny M, Cariou B, Meirhaeghe A, Di Filippo M. A new 165-SNP low-density lipoprotein cholesterol polygenic risk score based on next generation sequencing outperforms previously published scores in routine diagnostics of familial hypercholesterolemia. Transl Res. 2023 May;255:119-127. doi: 10.1016/j.trsl.2022.12.002. Epub 2022 Dec 15. PMID 36528340